CLINICAL TRIAL: NCT02343978
Title: Phase II, Randomized, Open-label Study of KWA-0711 Administrated Orally for 2 Weeks to Evaluate Its Safety and Efficacy in Patients With Chronic Constipation (CC)
Brief Title: Phase II Study of KWA-0711 in Patients With Chronic Constipation (CC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KWA1205
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; CC

ARMS (2):
- KWA-0711 High dose (Experimental)
  Interventions: Drug: KWA-0711
- KWA-0711 Low dose (Experimental)
  Interventions: Drug: KWA-0711

INTERVENTIONS:
Drug: KWA-0711

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of KWA-0711 in Chronic Constipation (CC) patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who experienced fewer than three Spontaneous Bowel Movements (SBMs) per week for more than 6 months prior to the enrollment
* The patients who experienced one or more of the following signs or symptoms during more than 25% of bowel movements for more than 6 months: straining, lumpy or hard stools, and a sensation of incomplete evacuation

Exclusion Criteria:

* Patients who have secondary constipation caused by systemic disorder
* Patients who have organic constipation
* Patients who received intestinal resection

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-12-26 (Actual); Primary Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 2 weeks

SECONDARY OUTCOMES:
Change in fasting and postprandial blood glucose levels | 2 weeks
Change in fasting and postprandial insulin levels | 2 weeks
ECGs, vital signs, and clinical labs | 2 weeks
Improvement of signs and symptoms associated with constipation | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Fukudo S, Endo Y, Hongo M, Nakajima A, Abe T, Kobayashi H, Nakata T, Nakajima T, Sameshima K, Kaku K; Mizagliflozin Study Group. Safety and efficacy of the sodium-glucose cotransporter 1 inhibitor mizagliflozin for functional constipation: a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Gastroenterol Hepatol. 2018 Sep;3(9):603-613. doi: 10.1016/S2468-1253(18)30165-1. Epub 2018 Jul 25. PMID 30056028